CLINICAL TRIAL: NCT06806111
Title: Wound Healing and Patient-Reported Outcomes After Autogenous Gingival Graft Harvesting from the Palate: a Randomized Controlled Clinical Trial
Brief Title: Wound Healing and Patient-Reported Outcomes After Gingival Graft Harvesting from the Palate
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Gonzalo Blasi, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER-ECL-2024-10
Record Dates: First submitted 2025-01-25; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Palatal Wound
Keywords: gingival graft harvesting; wound healing agent; postoperative pain; palatal healing; palatal volumetric changes
MeSH Terms: conditions — Pain, Postoperative | interventions — Sutures

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Suture (Active Comparator): This is the control group. In this group, 5-0 non-resorbable suspensory mattress sutures will be anchored to the soft tissues apical to the palatal wound area (5-0 Polypropylene, Prolene, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA).
  Interventions: Procedure: Suture
- Cyanoacrylate bioadhesive (Experimental): This is the test group. In this group, several drops of a high-viscosity cyanoacrylate bioadhesive will be applied (Cuantum Oral Adhesive, Cuantum Medical Cosmetics S.L., Spain) to create a uniform adhesive layer. No sutures will be placed.
  Interventions: Procedure: Cyanoacrylate bioadhesive

INTERVENTIONS:
Procedure: Suture — Hemostatic sutures at the palatal donor site; 5-0 non-resorbable suspensory mattress sutures will be anchored to the soft tissues apical to the palatal wound area (5-0 Polypropylene, Prolene, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA).
  Arms: Suture
Procedure: Cyanoacrylate bioadhesive — Several drops of a high-viscosity cyanoacrylate bioadhesive will be applied (Cuantum Oral Adhesive, Cuantum Medical Cosmetics S.L., Spain) to create a uniform adhesive layer.
  Arms: Cyanoacrylate bioadhesive

SUMMARY:
The goal of this clinical trial is to evaluate whether two different techniques for treating palatal wounds-sutures and cyanoacrylate bioadhesive-can influence postoperative morbidity, clinical healing, and soft tissue dimensional changes in patients undergoing epithelialized gingival graft harvesting from the palate. The main questions it aims to answer are:

Does the use of cyanoacrylate bioadhesive reduce postoperative morbidity compared to sutures? Does the choice of wound treatment technique affect clinical healing and three-dimensional changes in soft tissues? Researchers will compare the sutures (control group) to the cyanoacrylate bioadhesive (test group) to determine if the bioadhesive leads to improved postoperative outcomes.

Participants will:

Undergo epithelialized gingival graft harvesting from the palate. Receive either sutures or cyanoacrylate bioadhesive for wound closure. Be monitored for postoperative morbidity, clinical healing, and soft tissue dimensional changes.

DETAILED DESCRIPTION:
Objectives Overall objective The aim of this randomized controlled clinical trial is to evaluate the clinical, volumetric, and patient-centered outcomes of autogenous gingival graft harvesting when treating the palate with different protective agents.

Specific objectives

* To assess wound healing, volumetric changes, post-operative pain and bleeding, eating discomfort, and analgesic consumption after EGG harvesting and protecting the palate with the following agents: (1) suturing; (2) cyanoacrylate bioadhesive.
* To assess any correlations between palate wound healing dynamics and patient-reported outcomes.
* To determine which demographic, anatomical, and surgical factors are correlated with higher post-operative pain and discomfort.

Hypothesis Null hypotheses

* H01: Using different palate protection agents provides similar wound healing and patient-reported outcomes.
* H02: There are no correlations between palate wound healing dynamics and patient-reported outcomes.
* H03: There are no correlations between demographic, anatomical, and surgical factors with higher post-operative pain and discomfort.

Alternative hypotheses

* H11: The use of different palate protection agents provides different wound healing and patient-reported outcomes.
* H12: There is a correlation between palate wound healing dynamics and patient-reported outcomes.
* H13: There are correlations between demographic, anatomical, and surgical factors with higher post-operative pain and discomfort.

Materials and methods

* Study design This study will be designed as a randomized controlled clinical study with parallel arms and a 2-month postoperative follow-up period.
* Setting of the study The study will be performed at the university clinic (CUO) of Universitat Internacional de Catalunya of Barcelona, Spain (UIC). Subjects will be selected, on a consecutive basis, among individuals referred to the Department of Periodontology at UIC. The study protocol and informed consent was reviewed by the Ethical Committee of the Universitat Internacional de Catalunya, Barcelona, Spain, and will be conducted according to the Helsinki Declaration, 1975, as revised in 2013.
* Study population Patients requiring mucogingival surgery for root coverage or soft tissue augmentation will be recruited.
* Pre-surgical treatment For periodontal patients, steps 1 and 2 of periodontal therapy will be completed before surgery. All patients will receive pre-surgical prophylaxis and oral hygiene instructions.
* Surgical treatment and study groups The surgeries will be performed by the postgraduate students of the Master's Degree in Periodontology at UIC Barcelona, Spain. Patients will be randomly assigned to one of the two groups using a computer-generated randomization table. Each patient's assigned group will be communicated to the operator through a sealed envelope that will be opened during the surgery, immediately after the graft harvesting procedure is completed. On the day of the surgery, local anesthesia will be administered (4% Articaine with epinephrine 1:100,000), and an EGG will be harvested with a 15C blade. The dimensions of the graft will be decided by the surgeon, according to treatment needs. For bilaminar techniques, the harvested graft will be extra-orally de-epithelialized (DGG), while the epithelium will be maintained in cases utilizing free gingival graft techniques. After covering the palatal wound with sterile gauze for a few seconds, the wound will be treated according to the patient's randomized assigned procedure: (1) suturing; (2) cyanoacrylate bioadhesive.

  1. Suturing (Control Group) In this group, 5-0 non-resorbable suspensory mattress sutures will be anchored to the soft tissues apical to the palatal wound area (5-0 Polypropylene, Prolene, Ethicon, Johnson and Johnson, New Brunswick, NJ, USA).
  2. Cyanoacrylate bioadhesive (Test Group) In this group, several drops of a high-viscosity cyanoacrylate bioadhesive will be applied (Cuantum Oral Adhesive, Cuantum Medical Cosmetics S.L., Spain) to create a uniform adhesive layer. No sutures will be placed.
* Post-surgical instructions and infection control Patients will be instructed to avoid mechanical trauma or brushing in the surgical sites for 2 weeks. Analgesics (ibuprofen 600 mg t.i.d for 5 days) will be prescribed and patients will be instructed to rinse with Chlorhexidine 0.12% b.i.d. for two weeks when sutures are removed. After suture removal, patients will resume mechanical toothbrushing with a soft toothbrush.
* Blindness The two clinical examiners will not be aware of the treatment allocation. However, because of the study design (suture vs. no suture), during the first weeks maintaining blindness will be impossible. The researcher who will perform the digital measurements will be blinded. Blindness will be maintained strictly confidential by the investigators.
* Data collection A guidebook will be prepared to systematize the procedures for sample and data collection. The data will be later transferred to a computerized database (Epidata®, Odense, Denmark, Europe).
* Sociodemographic data An interview will be conducted during the pre-surgical visit to obtain information regarding age, gender, medical history, current medications, smoking habits, and previous periodontal surgeries.
* A questionnaire will be prepared and handed to patients on the day of the surgery. Patients will be instructed to answer the questions at the same time of the day and refer only to the palatal wound. Post-operative pain, post-operative bleeding, discomfort at eating, and analgesic consumption will be assessed. At the final follow-up visit (8 weeks), patients will be handed an Oral Health Impact Profile questionnaire (OHIP5) to assess the influence of the intervention on their quality of life.
* Clinical outcomes such as the graft dimensions and the Palatal Wound Healing Score will be evaluated.The palatal wound healing score will be assessed by two blinded clinical examiners independently. The inter-rater reliability will be calculated to validate the score.
* A digital dental scan of the whole arch will be taken with an intraoral scanner (3Shape Trios, Copenhagen, Denmark) using a bilateral mouth retractor to obtain standard tessellation language (STL) files. The acquired data will be transferred into digital imaging software (3Shape Trios®, Erlangen, Germany) in which the patient name will be substituted by a random ID number to anonymize the data. The STL model at baseline (T0) will be considered as a reference, and consecutively, the digital surface models after immediate EGG harvesting (T1), at 1-week postsurgery (T2), 2 weeks (T3), 3 weeks (T4), 4 weeks (T5), and 8 weeks (T6), will be imported and aligned using the "initial alignment" and "best-fit alignment" tools (Geomagic, 3D Systems, Research Triangle Park, NC, USA) using the tool Control X. To guarantee maximum accuracy, the palatal surfaces of the concerned teeth will be used as reference landmarks for the alignment of the different time points. The Region of Interest (ROI) will be determined as a rectangular shape corresponding to the palatal wound immediately after epithelial gingival graft harvesting. The digital measurements will be performed by a single, calibrated examiner. The intra-operator reliability will be measured on 10 random patients before the measurements of the study cases. The following measurements will be performed: the Wound Area, the mean distance between baseline and follow-up surfaces at the level of the Region Of Interest; linear Dimensional changes.
* A Cone Beam Computed Tomography (CBCT) will be performed before the surgery and the Digital Imaging and Communication in Medicine (DICOM) and STL of the immediate post-op will be superimposed using an implant planning program (Bluesky Bio). The following measurements will be taken: initial palatal thickness; remaining palatal thickness, measured in the center of the graft at the 3 levels mentioned above.
* Sample size calculation Based on a previous study, the sample size was calculated using post-operative pain as the primary outcome. Assuming a similar Standard Deviation (2.4) and effect size (f) of 0.81, a minimum of 50 patients is needed to detect a significant difference in pain levels with 80% power. To account for an estimated dropout rate of 20%, the sample size was adjusted to 66 patients. This will ensure adequate power to detect large effect sizes for graft area and Visual Analog Scale (VAS) pain scores. Therefore, 33 patients are deemed necessary in each group to achieve the significance level of 0.05.
* Statistical analysis Descriptive statistics will be performed for continuous and categorical variables using means and standard deviations or frequencies and percentages. The Kruskal-Wallis (continuous variables) or chi-square (categorical variables) tests will analyze characteristics across the treatment groups. Multiple random effects regression models will be applied to evaluate VAS changes across the three groups over time. Adjustments will be performed for gender, age, and clinical characteristics (graft height, width, and thickness). Group-time interaction will be tested using a global Wald test. Differences between baseline and post-operative follow-ups will be analyzed using the Wilcoxon test (quantitative variables) or paired t-student according to the distribution of the data and McNemar's test (qualitative variables). The association between Wound Healing Score and Wound Area from one hand and post-operative pain, post-operative bleeding, discomfort at eating, and analgesic consumption from the other hand, will be evaluated using the Mann-Whitney U test or the t-student, depending on the distribution of the data. To disclose associations between them, the Pearson or Spearman correlations will be employed. The level of statistical significance will be set at p < 0.05. Statistical analyses will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy individuals older than 18 years old;
* Healthy periodontal status according to the AAP/EFP definition;
* Full-mouth plaque (FMPS) and bleeding scores (FMBS) ≤ 20%;
* No history of soft tissue harvesting.

Exclusion Criteria:

* Pregnancy or lactation;
* Self-reported smoking ≥10 cigarettes/day;
* Metabolic diseases that negatively affect soft tissue healing (i.e., diabetes mellitus);
* Any medication that may interfere with wound healing;
* Removable maxillary prostheses;
* Ongoing orthodontic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain | 1 day, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks
  Minimum and maximum values [0-100] Higher scores mean worse outcome (more pain) A questionnaire will be prepared and handed to patients on the day of the surgery. Patients will be instructed to answer the questions at the same time of the day and refer only to the palatal wound.
  Postoperative pain will be assessed using a Visual Analog Score (VAS) at 1 day, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks postoperatively.

SECONDARY OUTCOMES:
Postoperative bleeding | 1 day, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks.
  YES/NO question, Yes meaning there is bleeding A questionnaire will be prepared and handed to patients on the day of the surgery. Patients will be instructed to answer the questions at the same time of the day and refer only to the palatal wound.
  Post-operative bleeding will be assessed dichotomously (YES/NO) at 1 day, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks.
Discomfort at eating | 1 day, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks
  Minimum and maximum values [0-100] Higher scores mean worse outcome (more discomfort) A questionnaire will be prepared and handed to patients on the day of the surgery. Patients will be instructed to answer the questions at the same time of the day and refer only to the palatal wound. Discomfort at eating will be assessed by using a VAS at 1 day, 3 days, 1 week, 2 weeks, 3 weeks, and 4 weeks postoperatively.
Analgesic consumption | during the first week
  Number of Ibuprofen pills taken during the first week postoperatively Higher number means worse outcome (more painkillers) A questionnaire will be prepared and handed to patients on the day of the surgery. Patients will be instructed to answer the questions at the same time of the day and refer only to the palatal wound. Analgesic consumption (n) will be reported during the first week postoperatively.
Oral Health Impact Profile 5 questionnaire (OHIP5) | At 8 weeks
  At the final follow-up visit (8 weeks), patients will be handed an Oral Health Impact Profile 5 questionnaire (OHIP5) to assess the influence of the intervention on their quality of life.
  The Spanish version of the validated OHIP5 consists of the following questions:
  Have you had difficulty biting food because of problems with your teeth, mouth, or dentures? Have you had painful discomfort in your mouth? Have you felt discomfort about the appearance of your teeth, mouth, or dentures? Have you noticed less taste in your food because of problems with your teeth, mouth, or dentures? Have you had difficulty doing your usual work because of problems with your teeth, mouth, or dentures? Responses will be marked on the following scale: 0-never; 1-hardly ever; 2 occasionally; 3-fairly often; and 4-very often.
Epithelial gingival graft dimensions | Per-operatively
  A periodontal probe (PCP UNC 15, Hu-Friedy, Chicago, IL, USA) will be used to measure the width, height, and thickness of the harvested graft in millimeters before de-epithelialization and fatty tissue removal.
Palatal Wound Healing Score | at 1 week, 2 weeks, 3 weeks, 4 weeks, and 8 weeks
  Minimum and maximum values [0-12] Higher scores mean better outcome (better healing) The palatal wound healing score will be assessed by two blinded clinical examiners independently at 1 week, 2 weeks, 3 weeks, 4 weeks, and 8 weeks. The inter-rater reliability will be calculated to validate the score.
  Variables 0 1 2 Necrosis: Complete; Incomplete; Absent Fibrin/granulation: tissue Fibrin > granulation tissue; Fibrin = granulation tissue; Fibrin < granulation tissue Bleeding on palpation: Present; Slight; Absent Epithelization: Absent; Incomplete; Complete Texture: Obvious difference; Moderate difference; No difference Scar tissue: Present; Slight; Absent
Wound Area | at 1 week, 2 weeks, 3 weeks, 4 weeks, and 8 weeks
  Measured in millimeters square The Wound Area; corresponding to the area of the ROI (WA in mm2). For this measurement, a PLY file will be created to be able to assess the area by color-matching.
The mean distance between baseline and follow-up surfaces at the level of the Region Of Interest | at 1 week, 2 weeks, 3 weeks, 4 weeks, and 8 weeks
  The mean distance between baseline and follow-up surfaces at the level of the Region Of Interest (ROI); the difference in mean thickness of the reconstructed volume in millimeters.
Linear Dimensional changes | at 1 week, 2 weeks, 3 weeks, 4 weeks, and 8 weeks
  Linear Dimensional changes; the mean palatal thickness change will be measured in 3 individually defined areas; the ROI will be divided into 4 equal parts by 3 vertical planes, and measurements will be made in the center of the graft at these 3 levels in millimeters.
Initial palatal thickness | Baseline
  A CBCT will be performed before the surgery and the Digital Imaging and Communication in Medicine (DICOM) and Standard Tesselation Language (STL) of the immediate post-op will be superimposed using an implant planning program (Bluesky Bio).
  The initial palatal thickness will measured in the center of the graft at the 3 levels mentioned above in millimeters.
Remaining palatal thickness | Immediate post-operative
  A CBCT will be performed before the surgery and the DICOM and STL of the immediate post-op will be superimposed using an implant planning program (Bluesky Bio).
  The remaining palatal thickness will be measured in the center of the graft at the 3 levels mentioned above in millimeters.

IPD SHARING:
Plan to Share IPD: Yes
The IPD to be shared will include:
  * Demographic data (e.g., age, gender, relevant medical history)
  * Clinical outcome measures, including postoperative morbidity, pain scores, and healing assessments
  * Three-dimensional soft tissue measurements, obtained from digital scans or clinical evaluations
  * Treatment allocation and intervention details, without identifiable information
Supporting Information: Study Protocol, CSR
Time Frame: After publishing
Access Criteria: Researchers must submit a formal data request outlining the purpose of their study, the specific data required, and the intended use.